CLINICAL TRIAL: NCT06330662
Title: Effectiveness of Hyaluronic Acid on Multiple Adjacent Gingival Recessions Using a Coronally Advanced Flap: Randomized Controlled Trial With One Year Follow-up
Brief Title: Effectiveness of Hyaluronic Acid on Multiple Adjacent Gingival Recessions Using a Coronally Advanced Flap
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Andelina Sekelja (Other)
Responsible Party: Sponsor-Investigator, Andelina Sekelja, doctor of dental medicine, University of Zagreb
Organization: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 05-PA-30-19-6/2023.
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Gingival Recession
Keywords: periodontal surgery; hyaluronic acid; coronally advanced flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: The control group refers to surgical intervention using a coronally advanced flap to cover multiple gingival recessions without the addition of hyaluronic acid (CAF) and the experimental group indicates the surgical intervention using a coronally advanced flap to cover multiple adjacent gingival recessions with the addition of hyaluronic acid intraoperatively (CAF + HA).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization would first be generated using a computer-selected program, and then the protocol itself would be placed in opaque sealed envelopes and handed to the operator immediately before the procedure with a decision as to whether or not hyaluronic acid (HA) would be applied. In treated areas where HA will not be applied, the operative site will be treated only with saline. The patient as well as the researcher and the outcomes assesssor will not be informed which patient belongs to which group. Randomization and allocation of envelopes as well as allocation of patients to groups will be determined by a fourth party.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coronally advanced flap with the hyaluronic acid (Experimental): The experimental group indicates the surgical intervention using a coronally advanced flap to cover multiple adjacent gingival recessions with the addition of hyaluronic acid intraoperatively (CAF+HA).
  Interventions: Procedure: Testing the effectiveness of hyaluronic acid in experimental group using a coronally advanced flap compared to a control group using a coronally advanced flap only
- Coronally advanced flap (Other): The control group refers to surgical intervention using a coronally advanced flap only to cover multiple gingival recessions without the addition of hyaluronic acid (CAF).
  Interventions: Procedure: Testing the effectiveness of hyaluronic acid in experimental group using a coronally advanced flap compared to a control group using a coronally advanced flap only

INTERVENTIONS:
Procedure: Testing the effectiveness of hyaluronic acid in experimental group using a coronally advanced flap compared to a control group using a coronally advanced flap only — The potential benefit of adding hyaluronic acid (HA) to the coronally advanced flap (CAF) operative technique to cover multiple adjacent recessions has not been sufficiently investigated. Improving aesthetics is one of the primary goals of root recession coverage periodontal surgery, and little is known about the same in multiple adjacent gingival recession coverage therapy. In patients with a sufficient amount (≥2 mm) of keratinized tissue, the coronally advanced flap (CAF) has been shown to be very effective in the treatment of multiple recessions, especially in terms of aesthetic results. The researchers concluded from a database search (Epistemonikos, Cochrane, Medline) that there is no evidence to support the use of HA + CAF to achieve greater root coverage in the treatment of multiple gingival recessions.

SUMMARY:
The goal of this clinical randomized trial is to examine the effectiveness of hyaluronic acid in treatment of multiple adjacent gingival recessions in 2 groups. Control group will be presented by using a coronally advanced flap only (CAF) and experimental group will be presented with addition of hyaluronic acid to a coronally advanced flap (CAF+HA). The main question it aims to answer is: is there any difference in the reduction of multiple gingival recessions between the control (CAF) and the test group (CAF + HA)? The research would be conducted on subjects referred for specialist treatment at the Department of Periodontology (Faculty of dental medicine, University of Zagreb). A record would be kept of all patients who underwent a detailed clinical examination, those who did not meet the criteria for inclusion in the study and those who refused to participate in it. Participants who meet the inclusion criteria will undergo a detailed clinical examination and if they agree to participate in the research, they will sign the informed form. During the pre-treatment, patients will receive instructions and a demonstration on proper maintenance of oral hygiene as well as a teeth cleaning. In addition to the informed form, they will fill out the OHIP-14 questionnaire, and the researcher will measure the periodontal indices at the very beginning before the operation, as well as the Schiff index. Patients will be photographed at the baseline as well as at follow-up examinations. The total number of subjects would be 42, or 21 patients in the 2 observed groups. The control group refers to surgical intervention using a coronally advanced flap to cover multiple gingival recessions without the addition of hyaluronic acid (CAF) and the experimental group indicates the surgical intervention using a coronally advanced flap to cover multiple adjacent gingival recessions with the addition of hyaluronic acid intraoperatively (CAF + HA).

DETAILED DESCRIPTION:
Gingival recession is defined as a shift of the gingival margin towards the apical side in relation to the cemento-enamel junction, and teeth with a thinner periodontal phenotype are considered more prone to the same occurrence (Jepsen et al., 2018). The coronally advanced flap surgical technique is used to cover root recessions of one or more teeth, if sufficient tissue is present to be mobilized. In 2000., Zucchelli and de Sanctis described the coronally advanced flap technique for covering multiple adjacent gingival recessions in one procedure, and it is applicable and used in clinical practice.

Hyaluronic acid (HA) is a biocompatible and non-immunogenic linear polysaccharide of high molecular mass present in periodontal tissue that has anti-inflammatory and bacteriostatic effects and promotes healing of the surrounding tissue. The potential benefit of adding hyaluronic acid (HA) to the coronally advanced flap (CAF) operative technique to cover multiple adjacent recessions has not been sufficiently investigated. Improving esthetics is one of the primary goals of root recession coverage surgery procedures, and little is known about the same in multiple adjacent gingival recession coverage therapy. In patients with a sufficient amount (≥2 mm) of keratinized tissue, the coronally advanced flap (CAF) has been shown to be very effective in the treatment of multiple recessions, especially in terms of aesthetic results (Chambrone et al., 2018; Pini-Prato et al., 2014.) . The authors concluded by searching databases (Epistemonikos, Cochrane, Medline) that there is no evidence supporting the use of HA + CAF to achieve greater root coverage in the treatment of multiple adjacent gingival recessions.

The aim of this study is to examine the clinical efficacy of HA in combination with CAF for the treatment of multiple gingival recessions in root coverage, width and thickness of keratinized gingiva, and patient-reported clinical outcomes compared to CAF alone as monotherapy.

Implications: It is important for clinicians to choose an adequate therapy in order to achieve the best possible aesthetic and functional result when covering multiple adjacent gingival recessions, reduce postoperative pain, but also ensure an adequate cost-benefit ratio for the patient.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* people without systemic diseases and chronic regular therapy
* non-smokers
* percentage of areas affected by plaque (FMPS) and percentage of bleeding sites on probing (FMBS) ≤25%
* the presence of a non-carious cervical lesion (NCCL) associated with recession
* gingival recessions on at least two adjacent teeth with a minimum depth of 2 mm and a clearly visible enamel-cement junction
* selection of patients capable of understanding and maintaining oral hygiene instructions with regular follow-up appointments
* selection of patients who fully understand the nature of the proposed surgical procedure and agree to informed consent

Exclusion Criteria:

* untreated periodontitis
* the presence of fixed prosthetic work (crown or bridge) on the examined adjacent teeth
* smokers
* pregnant and lactating women
* patients with uncontrolled type I and II diabetes
* patients with medical contraindications for surgical therapy
* medical history related to malignancies, radiotherapy, chemotherapy for the last 5 years
* taking chronic therapy that affects soft tissue healing such as: steroids, high doses of anti-inflammatory drugs, anticoagulants
* patients with active systemic infection
* allergies to hyaluronic acid
* allergies to local anesthesia
* alcohol or drug use
* participation in another clinical research in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
The effect of hyaluronic acid on recession reduction | 1 year
  The primary outcome is to examine the effectiveness of hyaluronic acid on the percentage of root coverage when treating multiple adjacent gingival recessions with the coronally advanced flap surgical technique

SECONDARY OUTCOMES:
To examine the effect of tissue thickness on recession coverage (KTt) | 1 year
  The thickness of the keratinized tissue will be measured intraoperatively at each teeth midline point from vestibular part of keratinized tissue during flap elevation using a digital caliper (Fervi® monoblock stainless steel electronic digital caliper Art. C041/150 0.01 mm)
To examine keratinized gingiva width (KTw) | 1 year
  The width of the keratinized gingiva will be measured intraorally using a periodontal probe (UNC 15, Hu Friedy®,Chicago IL, SAD) baseline and at follow-up examinations after 1 month, 3 months and 6 months postoperatively
To examine changes in periodontal clinical parameters: PPD | 1 year
  periodontal pocket probing depth (PPD) is the distance from the gingival margin to the apical portion of the gingival sulcus and will be measured at 3 points; mesial, buccal, distal part of the tooth using a periodontal probe (UNC 15, Hu Friedy®,Chicago IL, SAD) at baseline and follow-up examinations after 3 months and 6 months postoperatively
To examine changes in periodontal clinical parameters: CAL | 1 year
  clinical attachment level (CAL) is measured with the periodontal probe (UNC 15, Hu Friedy®,Chicago IL, SAD) as the distance from the cemento-enamel junction (CEJ) to the free gingival margin at baseline and follow-up examinations 3 months and 6 months postoperatively
To examine changes in periodontal clinical parameters: REC | 1 year
  Gingival recession is measured clinically as the distance from the cemento-enamel junction to the depth of the free gingival margin using the millimeter markings on the periodontal probe (UNC 15, Hu Friedy®,Chicago IL, SAD) baseline and at follow-up examinations after 1 month, 3 months and 6 months postoperatively
To examine changes in periodontal clinical parameters: FMPS (full mouth plaque score) | 1 year
  The presence of plaque will be measured at baseline and at follow-up examinations using a periodontal probe (UNC 15, Hu Friedy®, Chicago IL, USA) at 3 vestibular sites; mesial, buccal, distal. It is recorded using the value + or - and it is calculated afterwards as the number of tooth sites where plaque is recorded, divided by a total number of available sites multiplied by 100 (expressed as a percentage) baseline and at follow-up examinations after 1 month, 3 months and 6 months postoperatively
To examine changes in periodontal clinical parameters: FMBS (full mouth bleeding score) | 1 year
  The presence of bleeding sites will be measured at baseline and at follow-up examinations using a periodontal probe (UNC 15, Hu Friedy®, Chicago IL, USA) at 3 vestibular sites; mesial, buccal, distal after the PPD (periodontal pocket depth) measurements. Presence or absence of bleeding will be marked using a value of + or -. The number of sites where bleeding is recorded is divided by the total number of available sites in the mouth and multiplied by 100 to express the bleeding index as a percentage baseline and at follow-up examinations after 1 month, 3 months and 6 months postoperatively
Assess the healing quality of the operated area by using a RES scale | 1 year
  RES scale (eng. Root coverage esthetic score) in 5 categories;
  * changes evaluated based on the position of the gingival margin (GM); score 0,3,6
  * evaluation of marginal tissue contour changes (MTC); score 0 or 1
  * soft tissue texture evaluation (STT); score 0 or 1
  * evaluation of the alignment of the mucogingival junction (MGJ); score 0 or 1
  * gingival color evaluation (GC); score 0 or 1
Schiff test tooth examination | 1 year
  To assess tooth hypersensitivity (scale from 0 to 3) on vestibular surface of the tooth; It is determined by using an air stimulus from the dental unit in such way that the air is directed at an angle of 90 degrees to the vestibular surface of the tooth for 1 second duration from a distance of 1 centimeter. Adjacent teeth are protected with gloves on fingers. Score 0; the patient does not respond to the air stimulus, Score 1; the patient responds to the air stimulus but does not require interruption of the stimulus, Score 2; the patient reacts to the air stimulus and requires interruption or spontaneously withdraws from the stimulus, Score 3; the patient reacts to the stimulus, considers it painful and requests its termination.
To examine the impact of oral health on quality of life | 1 year
  Using the OHIP-14 questionnaire; it has been used to assess the impact of oral health problems on an individual's life. It consists of 14 questions, and patients complete it at baseline and at follow-up appointments 1 month, 3 months, 6 months postoperatively. Patients answer the offered 14 questions by circling the stated values: 0; never, 1; almost never, 2; occasionally, 3; often, 4; very often. OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. Higher OHIP-14 scores indicate worse, and lower scores indicate better OHRQol (Oral Health-related Quality of Life)
To evaluate the level of pain postoperatively during the healing of the surgical wound | 1 year
  By using the VAS scale and keeping a pain diary during the first 7 days postoperatively.
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a line with graphical display and two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). Patients will take the printed measurements scales with them at home and will be asked to mark pain intensity on the scale for the first seven days. Patients will also keep a pain diary where they will be asked to write the name of a painkiller they took, dosage, frequency of taking it and indication. The completed medication diary and the VAS scale are brought with them to the appointment 14 days after the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Zagreb - School of dental medicine, Zagreb, Hrvatska, Croatia

IPD SHARING:
Plan to Share IPD: No